CLINICAL TRIAL: NCT04984785
Title: Characterization of Physiological Mechanisms Involved in the Regulation of Eating Behavior for the Identification of Innovative Nutritional Strategies for Obese Patients Before and After Bariatric Surgery
Brief Title: Lipid Metabolism in Obese Subjects Undergoing Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Collaborators: Azienda Ospedaliera Brotzu (Other)
Responsible Party: Principal Investigator, Sebastiano Banni, Full Professor, University of Cagliari
Other Study IDs: unica
Record Dates: First submitted 2021-05-31; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Bariatric Surgery Candidate; Lipid Metabolism Disorders; Obesity
Keywords: Fatty Acids, Nonesterified; Peroxisome Proliferator-Activated Receptors; Endocannabinoids; N-acylethanolamines
MeSH Terms: conditions — Lipid Metabolism Disorders; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate modifications in the metabolism of polyunsaturated fatty acids (PUFA) and biosynthesis of the lipid mediators N-acylethanolamines (NAE), both known to induce and be induced by the nuclear peroxisome proliferator-activated receptor (PPAR)-α, which may also explain the well-established improved lipid and energy metabolism after bariatric surgery. The study is focused on understanding the weight loss mechanisms in order to develop targeted dietary protocols.

DETAILED DESCRIPTION:
The study involves a careful preliminary medical history of the patients, with physical examination, anthropometric parameters measurements and blood sampling for blood chemistry routine and evaluation of any adverse events to assess suitability for the study. The evening before bariatric surgery, one month and six months after bariatric surgery anthropometric parameters measurements, blood sampling for blood chemistry routine, inflammatory and lipid-metabolomic profile, and evaluation of any adverse events are performed. For the study samples are stored identified by a code to be analyzed anonymously. Study interruption criteria are: development of allergic reactions, ketonemia> 1.5 mmol/L, acute gout

ELIGIBILITY:
Inclusion Criteria:

* subjects with pathological obesity suitable for bariatric surgery
* Body Mass Index (BMI) range 35-59

Exclusion Criteria:

* established diagnoses of a major disease (e.g., diabetes or kidney disease)
* pregnancy or breastfeeding,
* food allergies,
* use of drugs that could affect lipid metabolism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients eligible for bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Modifications of Endocannabinoid and N-acylethanolamine plasma levels | 6 months
  These lipid derivatives are involved in control of energy expenditure and lipid metabolism and are measured by LC MS/MS and expressed as nmol/ml plasma
Weight loss as kg, and fat mass reduction as total kg and percent of body mass | 6 months
  Indicators of the success of the intervention
Changes in fatty acid plasma profile induced by bariatric surgery | 6 months
  Fatty acid profile affect lipid derivatives. Fatty acid are measured by LC and GC and expressed as nmol/ml plasma

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Banni, PhD, Principal Investigator — Università di Cagliari
Locations (1):
- Centro di Chirurgia Bariatrica dell'Azienda Ospedaliera G. Brotzu, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No